CLINICAL TRIAL: NCT02151448
Title: A Phase 1/2 Trial Evaluating αDC1 Vaccines Combined With Tumor-Selective Chemokine Modulation as Adjuvant Therapy After Surgical Resection of Peritoneal Surface Malignancies
Brief Title: αDC1 Vaccine + Chemokine Modulatory Regimen (CKM) as Adjuvant Treatment of Peritoneal Surface Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: David Bartlett (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor-Investigator, David Bartlett, MD, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-110; 5P01CA132714-05 (NIH); 12-110 (Other: University of Pittsburgh Cancer Institute)
Record Dates: First submitted 2014-05-28; First posted 2014-05-30 (Estimated); Results first posted 2020-01-28 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-07

CONDITIONS: Malignant Neoplasm of Pancreas Metastatic to Peritoneal Surface; Malignant Peritoneal Mesothelioma; Peritoneal Carcinomatosis
MeSH Terms: conditions — Peritoneal Neoplasms | interventions — lentiviral minigene vaccine of COVID-19 coronavirus; AlkB Homolog 2, Alpha-Ketoglutarate-Dependent Dioxygenase; Celecoxib; Interferon alpha-2; Introns; poly(I).poly(c12,U); Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccine + chemokine modulatory regimen (Experimental): Week 1 (at recovery from surgery; ≥ 6 weeks post-surgery)-Priming Vaccine dose; no chemokine modulation; 1 day: αDC1 vaccine; Oral celecoxib, 200 mg, before & after treatment on day of vaccination; Weeks 2-3 -Rest; Week 4 (target) - Booster C1; Mon: αDC1 vaccine;Tues - Fri: Systemic Chemokine Modulation Regimen. Oral celecoxib, 200 mg, BID on vaccination days & CKM. Celecoxib will be dced after CKM on Fri. Rintatolimod only administered on Wed & Fri.; Week 5-7 -Rest; Week 8 (target) -Booster C2; Monday: αDC1 vaccine. Oral celecoxib, 200 mg, BID on days of vaccination and CKM. Tues - Fri:Systemic Chemokine Modulation Regimen. Rintatolimod only administered on Wed & Fri. Celecoxib will be dced after CKM on Fri.; Week 9-11 -Rest; Week 12 (target) -Booster C3; Monday: αDC1 vaccine. Tues-Fri: Systemic Chemokine Modulation Regimen. Rintatolimod only administered on Wed & Fri. Oral celecoxib, 200 mg, BID, given on days of vaccination and CKM. Celecoxib will be discontinued after CKM on Fri.
  Interventions: Biological: DC vaccine; Drug: Celecoxib; Drug: Interferon Alfa-2b; Biological: rintatolimod

INTERVENTIONS:
Biological: DC vaccine — Administered on Monday of each cycle: 1 intranodal ultrasound-guided injection (target dose of 3 x 10e6 cells in 0.5 mL) + 1 intradermal injection (target dose of 3 x 10e6 cells in 0.5 mL)
  Other Names: Alpha-type-1 polarized dendritic cells; alpha DC1; αDC1
Drug: Celecoxib — Administered at 200 mg, once a day orally, starting the day of the first DC vaccine through week 4/cycle 2. Participants will not take celecoxib while receiving standard of care chemotherapy as instructed by their local oncologist. Celecoxib will continue starting week 20/cycle 3 and continue until the Friday of the last day of the CKM administration, cycle 4. Administered at 400 mg, 200 mg twice a day orally, on days participants receive vaccine and CKM.
  Other Names: Celebrex; Celebra; Onsenal
Drug: Interferon Alfa-2b — Intravenous infusion over 20 minutes: doses tested in Phase 1 portion (5, 10, or 20 MU/m2) will determine the Phase 2 dose. Administered on the Tuesday of each CKM cycle.
  Other Names: Interferon-α2b; Intron A; IFN-α2b; IFNα; IFN; NSC #377523
Biological: rintatolimod — Intravenous infusion of 200 mg on Wednesday and Friday only of the CKM regimen. The protocol allows for de-escalation to 100 mg if attributable adverse effects are observed.
  Other Names: PolyIC12U; Ampligen®; poly I: polyC12U; Polyinosinic:polycytidylic-polyuridylic acid; polyriboinosinic/polyribocytidylic (uridylic) acid

SUMMARY:
This trial is to determine the safest dose of a triple combination (chemokine modulatory regimen or CKM) of celecoxib, interferon alfa (IFN), and rintatolimod that can be given with a DC vaccine as treatment of peritoneal surface malignancies after standard of care surgery.

The first phase of this study will determine the safest dose of IFN that can be given in combination with celecoxib and rintatolimod along with a DC vaccine. The doses of celecoxib (400 mg) and rintatolimod (200 mg) will be consistent while the dose of IFN will be increased (5, 10, or 20 MU/m2) as participants are enrolled to the trial. The high dose of IFN in combination with celecoxib and rintatolimod will be used for the next phase of the clinical trial. After surgery, participants will receive 2 cycles of the investigational treatment.

The second phase of this study will test if the investigational treatment has any effects on peritoneal surface malignancies. The doses of the combination determined in the first phase will be used in this phase of the clinical trial. After surgery, participants will receive 2 cycles of the investigational treatment, followed by standard chemotherapy as determined by their oncologist, and then 2 more cycles of the investigational treatment.

DETAILED DESCRIPTION:
This trial will evaluate the safety and effectiveness of autologous alpha-type-1 polarized dendritic cell (alpha-DC1) vaccines (patients' autologous alpha-DC1s loaded with autologous tumor material), combined with a systemic chemokine modulation regimen [CKM; intravenous rintatolimod (TLR3 ligand, a derivative of Poly-I:C) + intravenous interferon-alfa + oral celecoxib] as adjuvant therapy, after cytoreductive surgery (CRS) and hyperthermic intraperitoneal chemotherapy (HIPEC), in patients with peritoneal surface malignancies (PSM), including but not limited to malignant peritoneal mesothelioma and peritoneal carcinomatosis (PC) of appendiceal and colorectal origin.

All patients judged to have peritoneal surface malignancy and considered able to be cytoreduced to Peritoneal Cancer Index (PCI) Completeness of Cytoreduction (CC) score of 1 or less will undergo CRS + HIPEC. Postoperative immunotherapy will start at least 4 weeks after CRS + HIPEC.

Immunotherapy regimen will include four cycles of intranodal (3M cells) and intradermal (3M cells) αDC1 vaccines. Each booster αDC1 vaccine dose (treatment cycles 2-4) will be followed by 4-days of systemic CKM, starting the day after vaccination (IFNα [dose-escalation: 5-20 MU/m2], intravenous [IV], once a day for 4 days; rintatolimod [short-half-life TLR3 ligand] 200 mg intravenous [IV], on Wednesday and Friday only of the CKM regimen; and celecoxib 200 mg, orally, twice a day for 4 days). In order to avoid overlap between experimental immunotherapy and potential adjuvant chemotherapy (which can be clinically indicated as a part of standard care in the subset of patients), the experimental treatments will be interrupted after cycles 1 and 2, to allow adjuvant chemotherapy that is done for each patient's clinical care, and is not a part of this research study. Whenever clinically indicated as a part of standard care, adjuvant chemotherapy may start at least 5 days after completion of the 2nd cycle of immunotherapy (first booster vaccine plus the first CKM). The 3rd cycle of immunotherapy may start at least 5 days after the completion of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically confirmed peritoneal surface malignancies, including but not limited to malignant peritoneal mesothelioma and peritoneal carcinomatosis (PC) from presumed appendiceal and colorectal primary tumors. Most patients will have received extensive prior treatments, due to the recurrent nature of PC. Prior therapies involve previous CRS, local and systemic chemotherapies. None of these prior treatments disqualifies the patient from receiving the protocol-mandated experimental treatment.
* Patients must be deemed able to undergo optimal cytoreductive surgery (CRS) defined as CC-score of 0 or 1 based on imaging.

Cytoreduction is defined as the burden of residual disease nodules left at the end of surgery (CC-0: no visible disease; CC-1: residual tumor nodules ≤ 2.5 mm in size; CC-2: residual tumor nodules 2.5 mm - 2.5 cm in size; CC-3: residual tumor nodules > 2.5 cm in size).

* Patients may be enrolled in the study regardless of prior chemotherapy regimens
* An ECOG performance status of 0, 1 or 2
* Age equal to 18 years or older
* Patients must be able to understand and be willing to sign a written informed consent document
* Able to swallow pills
* Must have normal organ and marrow function as defined below:

Platelet ≥ 75,000/µL Hemoglobin ≥ 9.0 g/dL Hematocrit ≥ 27.0% Absolute Neutrophil Count (ANC) ≥ 1500/µL WBC >2000/mm3 Creatinine < 1.5 x institutional upper limit of normal (ULN), OR Creatinine clearance ≥ 50 mL/min/1.73 m2 for patients with creatinine levels greater than 1.5 x ULN Total bilirubin ≤ 1.5 x ULN AST(SGOT) and ALT(SGPT) ≤ 2.5 X ULN

* Must be eligible for pheresis within 8 weeks of surgery
* Availability of sufficient number of tumor cells for cryopreservation and subsequent vaccine production
* Must have had HIPEC during surgery
* Must have a CC score of 0

Exclusion Criteria:

* Infection of tumor tissue with pathogens resistant to radiation and fungizone
* Patients on systemic immunosuppressive agents, including steroids. Patients who are able to be removed from immunosuppressives at least 5 days prior to the first vaccine will be considered eligible.
* Patients with active autoimmune disease or history of transplantation. Patients with indolent or chronic autoimmune disease not requiring steroid treatment are considered eligible.
* Patients who are pregnant or nursing
* Patients experiencing a cardiac events (acute coronary syndrome, myocardial infarction, or ischemia) within the 3 months prior to accrual
* Patients with a New York Heart Association classification of III or IV
* Prior allergic reaction or hypersensitivity to celecoxib or NSAIDs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2014-07; Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L Bartlett, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Hillman Cancer Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- α DC1 Vaccine + Chemokine Modulatory Regimen: Phase 1:
  α DC1 vaccine and
  Chemokine Modulatory Regimen:
  Celecoxib: Administered at 200 mg, once a day orally (T-TH) Rintatolimod: Intravenous infusion of 200 mg (Wed & and Fri, only) Interferon Alfa-2b: Intravenous infusion - 5 MU/m^2 or 20 MU/m^2 (T-Fri)
  Phase 2 α DC1 vaccine and
  Chemokine Modulatory Regimen:
  Celecoxib: Administered at 200 mg, once a day orally (T-TH) Rintatolimod: Intravenous infusion of 200 mg (Wed & and Fri, only) Interferon Alfa-2b: Intravenous infusion - 20 MU/m^2 (T-Fri)
Period: Phase 1
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Started | 9
Completed | 9
Not Completed | 0
Period: Phase 2
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Started | 55
Completed | 55
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Includes all Phase 1 and Phase 2 participants.
Groups:
- α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen: Phase 1:
  α DC1 vaccine and
  Chemokine Modulatory Regimen:
  Celecoxib: Administered at 200 mg, once a day orally (T-TH) Rintatolimod: Intravenous infusion of 200 mg (Wed & and Fri, only) Interferon Alfa-2b: Intravenous infusion - 5 MU/m^2 or 20 MU/m^2 (T-Fri)
  Phase 2:
  α DC1 vaccine and
  Chemokine Modulatory Regimen:
  Celecoxib: Administered at 200 mg, once a day orally (T-TH) Rintatolimod: Intravenous infusion of 200 mg (Wed & and Fri, only) Interferon Alfa-2b: Intravenous infusion - 20 MU/m^2 (T-Fri)
Arm/Group | α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen
Number analyzed (Participants) | 64
Age, Continuous [Median (Full Range); unit: years] | 53 [27 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 42
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 61
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase 2 Dose (RP2D) (Phase 1)
Description: Number of patients treated at each of the three possible dose levels of Interferon α (5 MU/m^2, 10 MU/m^2 or 20 MU/m^2) during the Phase 1 portion of the study.
Time Frame: Up to 24 weeks
Population: Only includes patients participating in the Phase 1 portion.
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1- αDC1 Vaccine +1 Cycle of Chemokine Modulatory Regimen: α DC1 vaccine and
  Chemokine Modulatory Regimen:
  Celecoxib: Administered at 200 mg, once a day orally (T-TH) Rintatolimod: Intravenous infusion of 200 mg (Wed & and Fri, only) Interferon α -2b: Intravenous infusion - 5 MU/m^2, 10 MU/m^2 or 20 MU/m^2 (T-Fri)
Arm/Group | Phase 1- αDC1 Vaccine +1 Cycle of Chemokine Modulatory Regimen
Number analyzed (Participants) | 9
Participants
  5 MU/M^2IFN alpha | 5
  10 MU/M^2 IFN alpha | 0
  20 MU/M^2IFN alpha (RP2D) | 4

2. Primary Outcome: Adverse Events Possibly, Probably or Definitely Related to Study Treatment
Description: Number of participants with adverse events (by Grade) that were possibly, probably or definitely related to the combined study immunotherapy regimen (αDC1 vaccines + CKM) per CTCAE v 4.0 (Common Terminology Criteria for Adverse Events).
Time Frame: Up to 24 weeks
Population: Patients treated with at least 1 course of α DC1 vaccine + 1 cycle of chemokine modulatory regimen who were evaluable for for completing surgery.
Measure: Count of Participants; unit: Participants
Groups:
- α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen: α DC1 Vaccine
  and
  Chemokine Modulatory Regimen:
  Celecoxib: Administered at 200 mg, once a day orally (T-TH) Rintatolimod: Intravenous infusion of 200 mg (Wed & and Fri, only) Interferon Alfa-2b: Intravenous infusion - 5 MU/m^2 or 20 MU/m^2 (T-Fri)
Arm/Group | α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen
Number analyzed (Participants) | 38
Participants
  Anemia : Grade 1-2 | 3
  Anemia : Grade 3-4 | 1
  Blurred vision : Grade 1-2 | 1
  Blurred vision : Grade 3-4 | 0
  Bruising : Grade 1-2 | 1
  Bruising : Grade 3-4 | 0
  Chills : Grade 1-2 | 34
  Chills : Grade 3-4 | 0
  Diarrhea : Grade 1-2 | 7
  Diarrhea : Grade 3-4 | 1
  Dizziness : Grade 1-2 | 1
  Dizziness : Grade 3-4 | 0
  Eye disorders - Other, specify : Grade 1-2 | 0
  Eye disorders - Other, specify : Grade 3-4 | 1
  Fatigue : Grade 1-2 | 15
  Fatigue : Grade 3-4 | 0
  Fever : Grade 1-2 | 7
  Fever : Grade 3-4 | 0
  Flu like symptoms : Grade 1-2 | 5
  Flu like symptoms : Grade 3-4 | 0
  Flushing : Grade 1-2 | 3
  Flushing : Grade 3-4 | 0
  General disorders and administration : Grade 1-2 | 7
  General disorders and administration: Grade 3-4 | 0
  Headache : Grade 1-2 | 10
  Headache : Grade 3-4 | 0
  Heart failure : Grade 1-2 | 0
  Heart failure : Grade 3-4 | 1
  Hypotension : Grade 1-2 | 1
  Hypotension : Grade 3-4 | 0
  Hypothyroidism : Grade 1-2 | 2
  Hypothyroidism : Grade 3-4 | 0
  Lymphocyte count decreased : Grade 1-2 | 4
  Lymphocyte count decreased : Grade 3-4 | 1
  Myalgia : Grade 1-2 | 3
  Myalgia : Grade 3-4 | 0
  Nausea : Grade 1-2 | 13
  Nausea : Grade 3-4 | 0
  Neutrophil count decreased : Grade 1-2 | 3
  Neutrophil count decreased : Grade 3-4 | 0
  Pain : Grade 1-2 | 6
  Pain : Grade 3-4 | 0
  Platelet count decreased : Grade 1-2 | 1
  Platelet count decreased : Grade 3-4 | 0
  Pleural effusion : Grade 1-2 | 1
  Pleural effusion : Grade 3-4 | 0
  Serum amylase increased : Grade 1-2 | 1
  Serum amylase increased : Grade 3-4 | 0
  Sinus bradycardia : Grade 1-2 | 2
  Sinus bradycardia : Grade 3-4 | 0
  Vomiting : Grade 1-2 | 7
  Vomiting : Grade 3-4 | 0
  Weight gain : Grade 1-2 | 1
  Weight gain : Grade 3-4 | 0
  White blood cell decreased : Grade 1-2 | 3
  White blood cell decreased : Grade 3-4 | 0

3. Secondary Outcome: Time to Progression (TTP)
Description: The length of time from the start of treatment until disease progression, per RECIST 1.1 considering only patients whose deaths were from cancer. Disease progression per RECIST 1.1 Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to18 months
Population: Patients treated with at least 1 course of α DC1 vaccine + 1 cycle of chemokine modulatory regimen who were evaluable for for completing surgery and response to treatment.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- α DC1 Vaccine + Chemokine Modulatory Regimen: α DC1 Vaccine
  and
  Chemokine Modulatory Regimen:
  Celecoxib: Administered at 200 mg, once a day orally (T-TH) Rintatolimod: Intravenous infusion of 200 mg (Wed & and Fri, only) Interferon Alfa-2b: Intravenous infusion - 5 MU/m^2 or 20 MU/m^2 (T-Fri)
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Number analyzed (Participants) | 55
months | 15.9 [13.6 to NA] — Upper bound not reached for 95% CI

4. Secondary Outcome: Overall Survival (OS)
Description: The length of time from the start of treatment that diagnosed patients are still alive.
Time Frame: Up to 5 years
Population: Patients treated with at least 1 course of α DC1 vaccine + 1 cycle of chemokine modulatory regimen who were evaluable for completing surgery.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Number analyzed (Participants) | 64
months | 52 [44 to NA] — Upper bound of 95% CI not reached.

5. Secondary Outcome: Progression-free Survival (PFS)
Description: The length of time during and after the treatment that patients remain alive with disease that does not progress. Per RECIST 1.1, Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
Time Frame: Up to 5 years
Population: Patients treated with at least 1 course of α DC1 vaccine + 1 cycle of chemokine modulatory regimen who were evaluable for completing surgery and response to treatment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Number analyzed (Participants) | 20
months
  colon cancer | 19 [9 to NA] — Upper bound not reached for 95% CI
  appendiceal cancer | 16 [14 to NA] — Upper bound not reached for 95% CI
  Mesothelioma | NA [NA to NA] — Median not reached.

6. Secondary Outcome: CXCL10 (Interferon Gamma-induced Protein 10) Levels
Description: Chemokine CXCL10 (Interferon gamma-induced protein 10) concentration levels measures in peripheral blood as a biomarker of anti-tumor activity. Increased levels can be predictive of good prognosis.
Time Frame: Prior to vaccine administration (Week 1), prior to vaccine booster (Week 4) and after vaccine booster (Week 8)
Population: Patients treated with at least 1 course of α DC1 vaccine + 1 cycle of chemokine modulatory regimen who were evaluable for completing surgery and response to treatment, and with ≥80% of samples available with measurable cytokine profiles via peripheral blood assay.
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Number analyzed (Participants) | 41
pg/mL
  Prior to vaccine administration (Week 1) | 1221.5 (135.4)
  Prior to vaccine booster (Week 4) | 16335.0 (59.3)
  After vaccine booster (Week 8) | 137.6 (17098.5)

7. Secondary Outcome: CXCL11 (C-X-C Motif Chemokine 11) Levels
Description: CXCL11 (C-X-C motif chemokine 11) protein concentration levels measures in peripheral blood. Increased levels can be predictive of good prognosis.
Time Frame: Prior to vaccine administration (Week 1), prior to vaccine booster (Week 4) and after vaccine booster (Week 8)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Number analyzed (Participants) | 41
pg/mL
  Prior to vaccine administration (Week 1) | 359.4 (340.2)
  Prior to vaccine booster (Week 4) | 12893.2 (190.3)
  After vaccine booster (Week 8) | 208.9 (5717.1)

8. Secondary Outcome: Interleukin 10 (IL-10) Levels
Description: Interleukin 10 (IL-10) (human cytokine synthesis inhibitory factor (CSIF)) concentration levels measures in peripheral blood. Increased levels of IL-10 is associated with advanced disease and poor prognosis.
Time Frame: Prior to vaccine administration (Week 1), prior to vaccine booster (Week 4) and after vaccine booster (Week 8)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/ml
Arm/Group | α DC1 Vaccine + Chemokine Modulatory Regimen
Number analyzed (Participants) | 41
pg/ml
  Prior to vaccine administration (Week 1) | 1.2 (2.4)
  Prior to vaccine booster (Week 4) | 7.9 (1.4)
  After vaccine booster (Week 8) | 7.5 (12.6)

9. Secondary Outcome: Interleukin 6 (IL-6) Cytokine Levels
Description: Interleukin 6 (IL-6) concentration levels measures in peripheral blood. Increased levels of IL-6 is associated with associated with advanced disease and poor prognosis.
Time Frame: Prior to vaccine administration (Week 1), prior to vaccine booster (Week 4) and after vaccine booster (Week 8)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen
Number analyzed (Participants) | 41
pg/mL
  Prior to vaccine administration (Week 1) | 15.2 (10.7)
  Prior to vaccine booster (Week 4) | 32.8 (19.0)
  After vaccine booster (Week 8) | 11.1 (32.7)

10. Secondary Outcome: Interleukin-8 (IL-8) Cytokine Levels
Description: Interleukin-8 (IL-8) cytokine concentration levels measures in peripheral blood. Increased levels of IL-8 is associated with associated with advanced disease and poor prognosis.
Time Frame: Prior to vaccine administration (Week 1), prior to vaccine booster (Week 4) and after vaccine booster (Week 8)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen
Number analyzed (Participants) | 41
pg/mL
  Prior to vaccine administration (Week 1) | 9.5 (15.7)
  Prior to vaccine booster (Week 4) | 16.9 (5.4)
  After vaccine booster (Week 8) | 28.6 (12.7)

11. Secondary Outcome: Stromal Derived Factor 1 Alpha (SDF-1A/CXCL-12) Chemokine Levels
Description: Levels of stromal derived factor 1 alpha (SDF-1A/CXCL-12) chemokine in peripheral blood. Higher levels of SDF-1A/CXCL-12 is associated with good prognosis.
Time Frame: Prior to vaccine administration (Week 1), prior to vaccine booster (Week 4) and after vaccine booster (Week 8)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen
Number analyzed (Participants) | 41
pg/mL
  Prior to vaccine administration (Week 1) | 1267.3 (5.0)
  Prior to vaccine booster (Week 4) | 2160.3 (476.8)
  After vaccine booster (Week 8) | 510.0 (852.2)

12. Secondary Outcome: Tumor Necrosis Factor (TFNα) Cytokine Levels
Description: Tumor necrosis factor (TFNα) cytokine concentration levels measures in peripheral blood. Higher TFNα levels is associated with good prognosis.
Time Frame: Prior to vaccine administration (Week 1), prior to vaccine booster (Week 4) and after vaccine booster (Week 8)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | α DC1 Vaccine + 1 Cycle of Chemokine Modulatory Regimen
Number analyzed (Participants) | 40
pg/mL
  Prior to vaccine administration (Week 1) | 10.8 (12.2)
  Prior to vaccine booster (Week 4) | 31.0 (5.0)
  After vaccine booster (Week 8) | 17.2 (25.4)

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Description: Adverse events data collected at screening, during clinical visit assessments and at follow-up and off treatment visits.
  Two Serious Adverse Events were Attributed to Study Treatment (2 events in 2 patients; excludes events from other causes):
  CARDIAC DISORDERS (Heart failure) EYE DISORDERS (Other)
Arm/Group | Vaccine + Chemokine Modulatory Regimen
All-Cause Mortality (participants affected / at risk) | 23/64
Serious Adverse Events (participants affected / at risk) | 17/64
Other Adverse Events (participants affected / at risk) | 46/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine + Chemokine Modulatory Regimen (N=64)
Heart failure (Cardiac disorders) | 1 — Attributed to Study Treatment
Eye disorders - Other, specify (Eye disorders) | 1 — Attributed to Study Treatment
Ileus (Gastrointestinal disorders) | 1 — Not Attributed to Study Treatment
Small intestinal obstruction (Gastrointestinal disorders) | 1 — Not Attributed to Study Treatment
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1 — Not Attributed to Study Treatment
Catheter related infection (Infections and infestations) | 1 — Not Attributed to Study Treatment
Infections and infestations - Other, specify (Infections and infestations) | 1 — Not Attributed to Study Treatment
Urinary tract infection (Infections and infestations) | 1 — Not Attributed to Study Treatment
Wound infection (Infections and infestations) | 1 — Not Attributed to Study Treatment
Alanine aminotransferase increased (Investigations) | 1 — Not Attributed to Study Treatment
Blood bilirubin increased (Investigations) | 1 — Not Attributed to Study Treatment
Lymphocyte count decreased (Investigations) | 1 — Not Attributed to Study Treatment
Neutrophil count decreased (Investigations) | 1 — Not Attributed to Study Treatment
White blood cell decreased (Investigations) | 1 — Not Attributed to Study Treatment
Hypokalemia (Metabolism and nutrition disorders) | 1 — Not Attributed to Study Treatment
Hyponatremia (Metabolism and nutrition disorders) | 1 — Not Attributed to Study Treatment
Flank pain (Musculoskeletal and connective tissue disorders) | 1 — Not Attributed to Study Treatment
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Not Attributed to Study Treatment
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Not Attributed to Study Treatment
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Not Attributed to Study Treatment
Thromboembolic event (Vascular disorders) | 1 — Not Attributed to Study Treatment
Colonic obstruction (Gastrointestinal disorders) | 2 — Not Attributed to Study Treatment
Diarrhea (Gastrointestinal disorders) | 2 — Not Attributed to Study Treatment
Serum amylase increased (Investigations) | 2 — Not Attributed to Study Treatment
Alkaline phosphatase increased (Investigations) | 3 — Not Attributed to Study Treatment
Hypertension (Vascular disorders) | 3 — Not Attributed to Study Treatment
Anemia (Blood and lymphatic system disorders) | 4 — Not Attributed to Study Treatment
Lipase increased (Investigations) | 4 — Not Attributed to Study Treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vaccine + Chemokine Modulatory Regimen (N=64)
Sinus bradycardia (Cardiac disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Weight gain (Investigations) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Flu like symptoms (General disorders) | 5
Blood bilirubin increased (Investigations) | 5
Creatinine increased (Investigations) | 5
Abdominal pain (Gastrointestinal disorders) | 6
Alanine aminotransferase increased (Investigations) | 6
Lipase increased (Investigations) | 7
Hypertension (Vascular disorders) | 7
General disorders and administration site conditions - Other, specify (General disorders) | 8
Pain (General disorders) | 8
Aspartate aminotransferase increased (Investigations) | 8
Platelet count decreased (Investigations) | 9
Vomiting (Gastrointestinal disorders) | 10
Alkaline phosphatase increased (Investigations) | 10
Serum amylase increased (Investigations) | 10
Lymphocyte count decreased (Investigations) | 11
Fever (General disorders) | 12
Neutrophil count decreased (Investigations) | 12
White blood cell decreased (Investigations) | 12
Hyponatremia (Metabolism and nutrition disorders) | 12
Diarrhea (Gastrointestinal disorders) | 14
Headache (Nervous system disorders) | 15
Hypoalbuminemia (Metabolism and nutrition disorders) | 16
Nausea (Gastrointestinal disorders) | 19
Fatigue (General disorders) | 19
Anemia (Blood and lymphatic system disorders) | 35
Chills (General disorders) | 36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-23): https://cdn.clinicaltrials.gov/large-docs/48/NCT02151448/Prot_SAP_000.pdf